CLINICAL TRIAL: NCT01589471
Title: The Value of Botox-A Administered as a Single Intra-rectal Injection for the Management of Low Anterior Resection Syndrome: A Phase II Study
Brief Title: The Value of Botox-A for Management of Low Anterior Resection Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE 11.088
Record Dates: First submitted 2012-04-27; First posted 2012-05-02 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2015-05

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer
Keywords: Low anterior resection syndrome; Botulinum toxin A; Quality of life; Incontinence; Rectal cancer; Anorectal manometry
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botox-A (Experimental): Intra-rectal (or intra-colic) injection of 100 U of Botox-A
  Interventions: Drug: intra-rectal Botulinum toxin A injection

INTERVENTIONS:
Drug: intra-rectal Botulinum toxin A injection — intra-colic injection of 100 U of Botulinum toxin A as a single injection distributed amongst the four quadrants, 5 cm above anastomosis
  Other Names: Botox (Allergan)

SUMMARY:
Low anterior resection syndrome (LARS) is frequent after treatment for low rectal cancer. Increased bowel frequency and urgency with rectal spasms and incontinence have deleterious impacts on quality of life in a third of the cases.

One possible physiopathology hypothesis suggests an ongoing spastic process; different mechanisms have been postulated. These include alteration of normal anorectal sensation with loss of the recto-anal inhibitory reflex (RAIR), decreased rectal compliance and reduced rectal capacity as well as sphincter damage secondary to preoperative chemoradiation therapy or during surgery.

Current available treatments are often ineffective, highlighting the need for more successful management. Botulinum toxin A (BTX-A) is a neurotoxin inhibiting acetylcholine release at the neuromuscular junction. It is currently used for the treatment of various smooth muscle spastic diseases.

The hypothesis of this study is that intra-rectal BTX-A injections could represent a medical treatment alternative for LARS. The goal of this study is to document the effects of intra-rectal BTX-A injections on sphincter function and quality of life of patients with LARS.

DETAILED DESCRIPTION:
No more information desired

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Aptitude to sign informed consent
* Diagnosis of low anterior resection syndrome (LARS) : More than 12 months after sphincter-preserving surgery for treatment of locally advanced rectal cancer, Mild to moderate underwear soiling, Baseline Wexner score ranging from 0-16 (moderate symptoms, and Patient-reported imperious defecation or Patient-reported incomplete stool evacuation
* Digital rectal exam (by surgeon) demonstrating satisfying anorectal tonus considering prior radical rectal surgery.
* Willingness to complete questionnaires and manometric studies before and after Botox-A administration
* Prior failed medical treatment, at least one attempt (narcotics, loperamide, cholestyramine, fibers)

Exclusion Criteria:

* Inability to sign informed consent
* Counter-indication to Botox-A administration : Allergy to Botox-A or its ingredients (Clostridium botulinum type A neurotoxin complex, human albumin and sodium chloride, Allergy to other forms of botulinum toxin (Dysport, Xeomin or Myobloc, Myasthenia gravis, Eaton-Lambert syndrome, lateral amyotrophic sclerosis or any other neurological disease which might interfere with neuromuscular function
* Prior use of any form of botulinum toxin A, for any indication
* Infection at proposed Botox-A injection site
* Personal or family history of bleeding diathesis
* Pregnancy or breastfeeding
* Severe incontinence (Wexner score ≥ 17 or daily use of diapers)
* Patient taking anticoagulant. ASA ( acetylsalicylic acid) allowed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of intra-rectal Botox-A injection on anorectal function as documented with standardized Wexner score | 1 month
Efficacy of intra-rectal Botox-A injection on anorectal function as documented with standardized Wexner score | 3 months

SECONDARY OUTCOMES:
Efficacy of intra-rectal Botox-A injection on anorectal function as documented with a visual scale for tenesmus and completeness of stool evacuation | 1 month and 3 months
Efficacy of intra-rectal Botox-A injection on quality of life as documented with EORTC-QlQ standardized questionnaires | 1 month and 3 months
  EORTC-QIQ is a quality of life questionnaire
Efficacy of intra-rectal Botox-A injection as documented with a patient medicine calender | 1 month
  patient-filled calender for usage of any medication intended for symptomatic treatment of LARS
Efficacy of intra-rectal Botox-A injection on anorectal function as documented with standardized anorectal manometry readings | 1 month
Long term efficacy of intra-rectal Botox-A injection on anorectal function as documented with Wexner score, EORTC-QLQ questionnaire and visual scale | 6 months
Safety of intra-rectal Botox-A injections as documented with adverse events monitoring | 1 month, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carole S Richard, MD FCRSC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada